CLINICAL TRIAL: NCT02044471
Title: The IMPULSE Pilot Study-- Investigating a Novel Synergy: Applying Ischemic Conditioning to Modulate the Altered Physiology From Contemporary continUous Flow Left Ventricular Assist Devices, to Reduce Stroke and Other Adverse Effects
Brief Title: The IMPULSE Study: Pilot
Acronym: IMPULSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Thoratec Corporation (Industry)
Responsible Party: Principal Investigator, Gilberto Defreitas, RN, Baylor College of Medicine
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: H-35006
Record Dates: First submitted 2014-01-21; First posted 2014-01-24 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Chronic Heart Failure
Keywords: left ventricular assist device; continuous flow; remote ischemic conditioning; hypertension; sympathetic tone; endothelial dysfunction
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Our intervention will be ischemic conditioning (IC) remotely applied using a sphygmomanometer. We will use the standard, validated protocol, which is inflation of the sphygmomanometer to 200 mmHg for 5 minutes, then deflation with 5 minutes of reperfusion, repeated for 3 cycles (total 30 minutes). This will be done in the dominant arm, twice daily.
  Once patients are discharged home on a stable pharmacotherapy regimen, they will be expected to follow the above intervention for 6 weeks, followed by another 6 weeks in the control (no intervention) phase. Patients will be randomized as to which phase they begin the study.
  Interventions: Other: Remote Ischemic Conditioning (using Sphygmomanometer)
- Control (No Intervention): standard care

INTERVENTIONS:
Other: Remote Ischemic Conditioning (using Sphygmomanometer) — Patients in experimental arm will have validated protocol of Remote Ischemic Conditioning (using Sphygmomanometer): 5 minutes with blood pressure cuff inflated at 200 mmHg, then deflated for 5 minutes; repeated for 3 cycles.
  Patient in control group will not perform this.
  Arms: Intervention

SUMMARY:
Continuous-flow (CF) left ventricular assist devices (LVADs) are an important tool in the treatment of end-stage heart failure, affording patients significantly improved quantity and quality of life. In recent years, tens of thousands of LVADs have been implanted worldwide, with nearly 1,000 at the Texas Heart Institute (THI). Despite the benefits from LVAD therapy, one major weakness is the high frequency of late strokes, reported up to 19%. CF LVADs minimize or remove the pulsatility within the blood system, introducing a new and incompletely understood physiology.

Increased sympathetic ("fight or flight" nervous system) tone secondary to lack of pulse in the blood system can cause high blood pressure, with subsequent hemorrhaging strokes (bleeding into the brain) are one possible explanation for this high adverse event rate in CF LVAD patients. A simple intervention to decrease the increased sympathetic tone is called "ischemic conditioning"; a sphygmomanometer (blood pressure cuff) is placed on the patient's arm to compress a major artery (ischemia) with subsequent release of the cuff (reperfusion) for set periods of time. This has been shown to reduce blood pressure and major adverse cardiovascular events in other patient populations.

We plan to conduct a trial to evaluate this intervention, ischemic conditioning, in patients with CF LVADs. We hypothesize that IC will cause a reduction in blood pressure and strokes in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* continuous flow LVAD and able to provide informed consent and comply with follow-up

Exclusion Criteria:

* < 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-08; Primary Completion 2016-04 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in mean doppler blood pressure | 6 weeks
  Patients will follow a standard, validated protocol for this non-invasive technique for 6 weeks, followed by 6 weeks in the control phase (or vice versa based on randomization of order). Each week, they will have Doppler blood pressure measurements and blood samples drawn for analysis.

SECONDARY OUTCOMES:
change in mean levels of inflammatory markers (TNFa, IL6, IL8, IL10) and endothelial function (adenosine, acetylcholine, bradykinin, nitric oxide, angiotensin, aldosternone) | 6 weeks
change in sympathetic neuronal activity | 6 weeks
  microneurographic measures of sympathetic function via peroneal nerve

CONTACTS AND LOCATIONS:
Overall Officials: Gilberto Defreitas, RN, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States